CLINICAL TRIAL: NCT05938868
Title: Efficacy of Low Intensity Pulsed Ultrasound and Low Level Laser Therapy on Osseointegration and Soft Tissue Healing Following Dental Implant Surgery: a Randomized Controlled Trial
Brief Title: Low Intensity Pulsed Ultrasound Versus Low Level Laser Therapy Post Dental Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Collaborators: Al Hayah University In Cairo (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/470001072023
Record Dates: First submitted 2023-07-01; First posted 2023-07-11 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Dental Implant; Surgical Dental Prostheses; Dental Implantation
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (LIPUS group) (Experimental): This group will include 17 patients who received Dental Implant Surgery. Patients will be treated with low intensity pulsed ultrasound in addition to standard care.
  Interventions: Device: Low intensity pulsed ultrasound (LIPUS); Other: Standard Care
- Group B (LLLT group) (Experimental): This group will include 17 patients who received Dental Implant Surgery. The patients will be irradiated with low level diode laser therapy (GaAs) in addition to standard care.
  Interventions: Device: low level diode laser therapy; Other: Standard Care
- Group C (Control group) (Active Comparator): This group will include 17 patients who received Dental Implant Surgery. Patients will be treated with standard care only after surgery for 2 weeks.
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: Low intensity pulsed ultrasound (LIPUS) — LIPUS will be delivered intra-orally using a probe applied on the buccal aspect of the implant site. The probe is in contact with the buccal attached gingiva with a thin film of intra oral gel intervening between them, acting as a transmitting medium. It will be applied twice a week for 20 minutes each session that commenced after surgery on the second day and continued for 10 weeks. The intensity of ultrasound therapy used was 30 mW/cm2 with a frequency of 1.5 MHz and temporal average power of 20 Mw
  Arms: Group A (LIPUS group)
Device: low level diode laser therapy — The patients will be irradiated with low level diode laser therapy (GaAs) (Chattanooga, model 27841, USA) .Patient will be irradiated with low level diode laser therapy with parameters: wavelength 850 nm and power of 200 mw in continuous mode will be applied in six points in non-contact method 10 mm away from the peri-implant soft tissue after suturing. The laser irradiations will be administered at six sites that included mesiobuccally, distobuccal, midbuccal, midlingual, mesial, and distal areas around implant for a duration of 10 seconds for each site. The total energy delivered was 6 J per session. And is based on a previous study by Gulati et al., 2020
  Arms: Group B (LLLT group)
Other: Standard Care — Patients in all three groups will receive the standard care which includes: (1) Extra-oral ice packs during the first 2 days every two hour; (2) maintain daily routine oral hygiene after surgery; (3) Patients will be instructed to eat a soft diet for one weeks; (4) Broad spectrum oral antibiotics in a dose of one capsule every twelve hours for a week; (5) Non-steroidal anti-inflammatory drugs at a dose of one tablet every 8 hours for four days; (6) Warm chlorhexidine gluconate solution as a mouthwash for a period of 2 weeks to enhance plaque control.

SUMMARY:
The purpose of the study is to investigate the significance difference between low intensity pulsed ultrasound (LIPUS) versus low-level laser therapy (LLLT) on osseointegration, soft tissue healing, pain pressure threshold and oral health related quality of life in patients post dental implant surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patients.
2. Both sexes will be contributed in the study.
3. Non-smokers.
4. Patients who needed dental implant in the maxillary or in the mandible.
5. Bone height and width no less than Class III bone quality assessed clinically and radiologically.

Exclusion Criteria:

1. Medically compromised patients as Uncontrolled diabetes mellitus.
2. Patients indicated for bone graft at the implant site.
3. Patients under chemotherapy or radiotherapy in facial region.
4. Poor oral hygiene.
5. Patients with any history of temporomandibular joint disorders.
6. Patients with any other periodontal and oral surgeries

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Changes in Osseointegration | Changes in Osseintegration immediately postoperative, after 6 weeks and after 3 months
  X-ray Radiograph will be performed for each patients and then analyzied by Specialized software to evaluate the osseointegration between bone and implant surface. The radiographs will be taken in high-resolution mode (Vista Scan Durr Dental, Durr Dental Italy S.r.l) with a dental X-ray machine (TM 2002 Planmeca Proline CC, Planmeca Group Helsinki, Finland) equipped with a long tube that operated at 70 Kw/7.5 mA. Specialized software (DBSWIN software, Durr Dental Italy S.r.l) will be used for linear measurements of marginal bone changes
Changes in soft tissue healing | Changes in soft tissue healing immediately postoperative, after 6 weeks and after 3 months
  Landry index for soft tissue healing will be used to measure soft tissue healing. The healing index (HI) evaluates healing based on redness, presence of granulation tissues, bleeding, suppuration, and epithelialization. A score of 1-5 was given with score 1 for very poor healing and 5 being excellent healing of the tissues. Higher scores indicate better healing rates. This index assesses the surgical wound by clinical examination.

SECONDARY OUTCOMES:
Changes in Pain pressure threshold | Changes in Pain pressure threshold immediately postoperative, after 6 weeks and after 3 months
  Pain pressure threshold at temporalis and masseter muscles will be measured at immediately post dental implant, after 6 weeks and after 3 months of treatment. A blinded assessor will use an algometer (FPX 25, Wagner Instruments, Greenwich CT, USA), a device that measures pressure or applied force on any part of the body, to register the pressure pain threshold (PPT) for temporalis and masseter muscles
Changes in oral quality of life | Changes in oral quality of life immediately postoperative, after 6 weeks and after 3 months
  Oral health-related quality of life is an established and relevant instrument with which to describe patient satisfaction. It will be measured at immediately post dental implant, after 6 weeks and after 3 months of treatment. OHRQoL consisting of 12-Item short-form Oral Health-Related Quality of Life Measures with a scale from 0 to 4 (Never, hardly ever, Occasionally, Fairly Often and Very Often) with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Abd El-Baky, Ph.d, Study Chair — Cairo University; Osama Gouda, Ph.D, Study Director — Faculty of Dentistry, Badr University; Hussein Mogahed, Ph.D, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahmoud ES, El-Baky AMA, Gouda OM, Hussein HG. Low intensity pulsed ultrasound versus low-level laser therapy on peri-implant marginal bone preservation and soft tissue healing following dental implant surgery: a randomized controlled trial. Head Face Med. 2025 Apr 23;21(1):29. doi: 10.1186/s13005-025-00502-z. PMID 40269949